CLINICAL TRIAL: NCT02797925
Title: Mechanisms Behind Development of Tendinopathy: Early Structural, Inflammatory, Nociceptive and Clinical Changes in Recreational Runners
Brief Title: Mechanisms Behind Development of Tendinopathy
Acronym: TESINaC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Peter Hung Thanh Tran, Doctor, phd student, Bispebjerg Hospital
Other Study IDs: BBH-128
Record Dates: First submitted 2016-06-02; First posted 2016-06-14 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Tendinopathy
Keywords: Achilles tendon; Patella tendon; Inflammation; Edema; Clinical; Structural
MeSH Terms: conditions — Tendinopathy; Inflammation; Edema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma and tissue.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Tendinopathy: Long slow strength training for 3 months that are performed at home or gym. Participants receive initial guidance to the exercises from a physiotherapist assigned to Bispebjerg H.
  Interventions: Other: Training
- Healthy: No intervention. No training

INTERVENTIONS:
Other: Training — Long slow strength training of the tendon for 3 months to improve function
  Other Names: Long slow strength training
  Groups: Tendinopathy

SUMMARY:
There has been an increasing amount of musculoskeletal injuries the past decades and overused tendons represents a major problem both for leisure and occupational activities. A full understanding of the pathophysiology of tendinopathy is very sparse and especially the early events in tendinopathy remains unexplained. In this phd study the investigators will investigate early changes in tendon tissue overloading and development of tendinopathy. The investigators will investigate sports-active individuals with recently developed tendinopathy with regards to symptoms (pain, function), tendon morphology (ultrasonography, MRI and electron microscopy), tendon mechanical properties (ultrasonography strain), tissue molecular biology (expression and content of matrix proteins), inflammation (activity of inflammatory pathways) and vascularization (Doppler and contrast enhancement US). The investigators hypothesize a coupling between early symptoms and inflammatory activity, followed by structural changes and altered mechanical properties. The investigation will indicate what symptoms and what tendon related determined measurements are primary for disease development ("tendinopathy blue prints") and should be regarding vital in prevention of tendinopathy.

DETAILED DESCRIPTION:
The investigators intend to study the development of tendinopathy in humans that enter a phase of relative overloading of their tendons. This will be done in a large cohort of individuals from whom the investigators have obtained basic data and tests. A percentage of these participants will develop overuse symptoms and in those the investigators will perform investigations that will identify the initial pathological changes in tendinopathy

Participants are included as soon as possible after diagnosis of either Achilles or patella tendinopathy because the investigators wish to investigate the early changes in tendinopathy. The hypothesis is, that at the early development of tendinopathy there will be a mismatch between matrix protein anabolic and catabolic pathways, and will be associated with a secondary upregulation of inflammatory and apoptotic markers in the tendon and result in hypervascularization and hyper-metabolism.

Recruiting participants will be done in collaboration with local athletic clubs in the Copenhagen area. The athletic clubs include Sparta, Københavns Idræt Forening (KIF), Frederiksberg Idræt Forening (FIF). Furthermore, the investigators will establish contact through online social media such as Facebook, Twitter and Google. In addition, Information leaflets will be handed out, and medical staff at the emergency rooms repeatedly informed about the project. Healthy participants can be directly recruited by participants already in the project, social medias and through information leaflets handed out. It is planned to inform staff at the emergency rooms at Bispebjerg Hospital, Amager Hospital, Gentofte Hospital, Herlev Hospital and Hvidovre Hospital. Patients and healthy controls can contact the primary investigator directly through email or telephone.

Recruitment to project TESINaC will focus onset of exercise pain and every participant will be evaluated by a doctor if the participant have tendinopathy or not. Once included the participant will undergo following procedures as soon as possible after diagnosis is given:

* Questionnaire regarding training history and ongoing symptoms
* Ultrasound scanning of tendons
* Ultrasound isometric
* Blood samples
* MRI of tendons on both legs MRI precedes biopsy as it can identify any diseased area within the tendon from which a biopsy can be taken. Only participants with tendinopathy will have to undergo biopsy from both patella tendons once during the project. Healthy participants will not undergo biopsy. No biopsy will be taken from the Achilles tendon as this procedure may worsen the participants symptoms.

Participants with tendinopaty will get physical reevaluated after 3, 6 and 12 months as regards to symptoms, activity of daily life, blood samples, questionnaires VISA-A/P and ultrasound measurements. Rehabilitation training of patients is expected to start as soon as possible after the biopsy have been taken.

Healthy participants will not be reevaluated nor will they undergo rehabilitation training.

It is expected that the results from this study will provide insight into the events leading up to a developing tendinopati. This study will add important information to understand the pathophysiology and provide information on timing of the phases as well. Information and results from the study will give insight into better treatment options that is more specific and earlier intervention on the individual basis. Furthermore, this study will investigate and address the question why some people develop tendinopathies and others do not when the training volume is equally raised.

ELIGIBILITY:
Inclusion Criteria:

* Marked tendon related pain in association with exercise on one leg
* Soreness during physical examination of patella or/and Achilles tendon upon palpation
* Demonstrate an ultrasonographic (US) thickening of the tendon (2 mm larger on the affected side vs the contralateral un-symptomatic side in the anterior-posterior projection)

Exclusion Criteria:

* Surgery in Achilles and/or patella tendon
* History of Achilles and/or patella tendinopathy
* Received any form of injection in Achilles and/or patella tendon
* Lately have infection around Achilles and/or patella tendon

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physical active participants over 18 years old, both men and women. The term physical active refers to any kind of sport and not only running. Participants with pain in either Achilles or patellar tendon on one leg. Healthy participants must be symptom free and not have any diseases at all.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Investigate the timespan of inflammation from acute phase to resolution in tendinopathy | 3 months
  Markers for inflammation includes tendon thickness, vascularization, inflammatory mRNA leves, inflammatory protein signals and mechanical properties of tendon.

SECONDARY OUTCOMES:
Measure tendon thickness in mm (anterior-posterior) on ultrasound | 3 months
Measure TNF-alpha mRNA levels in patella biopsies as ratio to GAPDH | 3 months
  GAPDH is a household gene and therefore expected to have constant mRNA levels. TNF-alpha mRNA is measured relative to GAPDH.
Measure the tendon region with maximal vascularization on ultrasound doppler signal based on visual impression from the investigators | 3 months
  The region with maximal vascularization is based on where the ultrasound doppler signal is most abundant, which depends on visual impression from the investigators.
IHC stain for TNF-alpha protein signal in patella biopsies with specific antibodies | 3 month
  Quantification is made by visual inspection of stained tendon samples
Measure tendon mechanical properties with ultrasound isometric | 3 months
  Tracking software provide details about deformation of tendon in mm, young modulus, max % strain and stiffness.
Measure CRP levels in blood samples | 3 months
  Systemic inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kjær, Professor, Study Director — Clinical Medicine
Locations (1):
- Bispebjerg Hospital, Copenhagen, Kbh NV, Denmark

IPD SHARING:
Plan to Share IPD: No